CLINICAL TRIAL: NCT05549050
Title: Correlation Between Interdialytic Weight Gain and Cardiovascular Diseases in Children With End-Stage Kidney Disease Undergoing Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Henny Adriani Puspitasari, Consultant of Pediatric Nephrology, Indonesia University
Other Study IDs: 21-10-1072
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: interdialytic weight gain; cardiovascular; chronic kidney disease; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: interdialytic weight gain — interdialytic weight gain during hemodialysis

SUMMARY:
This study aimed to discuss the correlation between interdialytic weight gain and cardiovascular diseases in children with end-stage kidney disease undergoing chronic hemodialysis. The cardiovascular parameters used include left ventricular hypertrophy, systolic and diastolic function, carotid intima-media thickness, myocardial circumferential strain, and strain rate.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease (chronic kidney disease stage 5)
* Undergo hemodialysis at least twice a week

Exclusion Criteria:

* History of congenital heart disease
* Critically ill patients with unstable hemodynamic status

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: End-stage kidney disease children aged 2-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between interdialytic weight gain and cardiovascular diseases in children with end-stage kidney disease undergoing hemodialysis | Through study completion, an average of 1 year
  Correlation between interdialytic weight gain and cardiovascular diseases in children with end-stage kidney disease undergoing hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Henny A Puspitasari, dr. Sp.A(K), Principal Investigator — Department of Child Health, Faculty of Medicine, University of Indonesia - Cipto Mangunkusumo Hospital
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided